CLINICAL TRIAL: NCT00064766
Title: A Prospective Randomized Clinical Trial of Doxycycline 20mg Twice a Day Versus Placebo on the Bleeding and Spotting in Women After Insertion of a Levonorgestrel Implant (Norplant) Protocol #2002-1
Brief Title: Norplant and Irregular Bleeding/Spotting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01HD043175 (NIH); NIH 1 R01 HD43175-01
Record Dates: First submitted 2003-07-11; First posted 2003-07-15 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Endometrial Bleeding; Periodontal Disease
Keywords: Norplant; Periodontal disease; Endometrial bleeding; Progestin-induced endometrial bleeding
MeSH Terms: conditions — Periodontal Diseases | interventions — Doxycycline

INTERVENTIONS:
Drug: doxycycline

SUMMARY:
Irregular or prolonged menstrual bleeding and/or spotting are common side effects in patients using progestin-only hormonal contraception such as levonorgestrel implants (Norplant). Doxycycline, a drug approved by the Food and Drug Administration (FDA) to treat gum disease, may reduce the occurrence of uterine bleeding and spotting in women who use Norplant. This study will evaluate the effects of doxycycline on uterine bleeding/spotting in women using Norplant.

DETAILED DESCRIPTION:
A high percentage of women using progestin-only contraception experience breakthrough bleeding (BTB) and spotting that causes impaired lifestyle and results in decreased compliance with this contraceptive method. There is a need for an effective, low-cost, easily adapted treatment to reduce the bleeding and spotting in progestin-only contraceptives. The molecular environment of the endometrium of women with BTB and spotting contains abnormally high levels of pro-inflammatory cytokines (TNF-alpha and IL-1 beta) and abnormally high levels of proteases (matrix metalloproteinases [MMPs] and neutrophil elastase), which prevent normal tissue repair. Doxycycline (DOX) is an inexpensive, FDA approved antibiotic that inhibits MMPs and reduces nitric oxide synthesis. This study will evaluate DOX treatment of progestin-only contraceptive induced BTB and spotting, characterize the endometrial molecular biologic changes that occur in DOX treated patients, and determine the effect of Norplant on sexual functioning and testosterone levels.

All participants in this study will receive Norplant. Participants will then be randomized to receive either DOX (20 mg twice a day) or placebo for 6 months. Participants will have 9 study visits during the 24 weeks of the study. Study visits will include a medical history, physical exam, and blood and urine tests. Participants will also have three periodontal evaluations and three endometrial biopsies. At the end of the study, participants may choose to have the Norplant implant removed if they wish to discontinue Norplant use; otherwise the implant may remain in for up to 5 years.

ELIGIBILITY:
Inclusion Criteria

* Regular menstrual periods for the last 2 cycles
* Currently not using hormonal contraceptives, including oral contraceptives, patch, ring, or Norplant in 2 months prior to study entry, or Depo-Provera in 12 months prior to study entry
* Currently not using tetracycline-class antibiotics
* Normal Pap smear

Exclusion criteria

* Pregnancy or breastfeeding within 2 months of study entry
* Chronic migraine headaches
* Uncontrolled high blood pressure
* Untreated sexually transmitted diseases
* Alcoholism or drug abuse within 12 months of study entry
* Insulin dependent diabetes
* Liver, kidney, or gallbladder disease
* Participation in another clinical trial within 30 days of study entry
* History of cancer
* History of blood clots, strokes, or heart disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2003-02; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: David F Archer, MD, Principal Investigator — CONRAD Clinical Research Center, Eastern Virginia Medical School
Locations (1):
- CONRAD Clinical Research Center, Eastern Virginia Medical School, Norfolk, Virginia, United States